CLINICAL TRIAL: NCT00452426
Title: Multi-center Pivotal Clinical Trial to Compare the Safety and Effectiveness of Procedural Sedation in GI Endoscopy: A Computer-Assisted Personalized Sedation (CAPS) Device Versus Current Standard of Care
Brief Title: Safety and Effectiveness of a Computer-Assisted Personalized Sedation (CAPS) Device for Propofol Delivery During Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: James Martin, EES
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CI-06-0004
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-12

CONDITIONS: Colonoscopy; Endoscopy, Digestive System; Conscious Sedation
Keywords: Propofol; Diprivan; Colonoscopy; Endoscopy, Digestive System; Conscious Sedation
MeSH Terms: interventions — Benzodiazepines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedation System (Experimental): Computer-Assisted Personalized Sedation (CAPS) device used for delivery of sedation
  Interventions: Device: Computer-Assisted Personalized Sedation (CAPS) Device (SEDASYS® System)
- Current Standard of Care (Active Comparator): Site's current standard used for delivery of sedation
  Interventions: Other: benzodiazepines and opioid sedation

INTERVENTIONS:
Device: Computer-Assisted Personalized Sedation (CAPS) Device (SEDASYS® System) — propofol sedation per device instructions for use
  Arms: Sedation System
Other: benzodiazepines and opioid sedation — per site's current standard of care
  Arms: Current Standard of Care

SUMMARY:
Patients routinely receive sedation during a colonoscopy or upper endoscopy (esophagogastroduodenoscopy; EGD) procedure. Propofol is a sedative that can be used during these procedures. The purpose of this study is to determine if this CAPS device enables a physician/registered nurse (RN) team to safely and effectively administer propofol sedation during colonoscopy or EGD procedures relative to current sedation practices.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Able to comprehend, sign, and date the written informed consent form
* English as primary language
* Undergoing a non-emergent EGD or colonoscopy
* Have taken nothing by mouth for a minimum of 6 hours prior to the study procedure
* American Society of Anesthesiologists (ASA) Class I, II or III

Exclusion Criteria:

* Allergy or inability to tolerate study medications or components of study medications
* Investigator anticipates greater than 45 minute procedure time due to known anatomical difficulty
* Currently using a fentanyl patch
* History of diagnosed sleep apnea
* History of diagnosed gastroparesis
* Baseline oxygen saturation < 90% (room air)
* Pregnant or nursing females
* Body mass index (BMI) ≥ 35
* Participation in a clinical trial within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Martin, PhD, Study Director — Ethicon Endo-Surgery, Inc.
Locations (7):
- United States (7):
  - Metropolitan Gastroenterology Group, PC, Washington D.C., District of Columbia
  - Fayetteville Gastroenterology Associates, PA, Fayetteville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Digestive Health Specialists, Tacoma, Washington

REFERENCES:
- [Derived] Pambianco DJ, Vargo JJ, Pruitt RE, Hardi R, Martin JF. Computer-assisted personalized sedation for upper endoscopy and colonoscopy: a comparative, multicenter randomized study. Gastrointest Endosc. 2011 Apr;73(4):765-72. doi: 10.1016/j.gie.2010.10.031. Epub 2010 Dec 18. PMID 21168841

RESULTS

PARTICIPANT FLOW:
Groups:
- Sedation System: Computer-Assisted Personalized Sedation (CAPS)device used for delivery of sedation
Period: Overall Study
Arm/Group | Sedation System | Current Standard of Care
Started | 496 | 504
Completed | 489 | 493
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedation System | Current Standard of Care | Total
Number analyzed (Participants) | 496 | 504 | 1000
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (13) | 53 (14) | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 248 | 514
  Male | 230 | 256 | 486
Region of Enrollment [Number; unit: participants]
  United States | 496 | 504 | 1000

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Oxygen Desaturation (AUCDesat)
Description: AUCDesat measures desaturation as a function of incidence, magnitude, and duration. AUCDesat is the difference between the threshold and actual oxygen saturation measured every second. The total area below the 90% threshold is summated to determine AUCDesat in units of seconds*percent.
Time Frame: From administration of initial drug dose until subject recovered from effects of sedation
Population: This analysis was intention to treat (ITT) which is all subjects who enrolled and had data avaiable. The differences in total subjects enrolled and subjects analyzed are due to missing data.
Measure: Mean (95% Confidence Interval); unit: seconds*percent of oxygen desaturation
Arm/Group | Sedation System | Current Standard of Care
Number analyzed (Participants) | 491 | 486
seconds*percent of oxygen desaturation | 23.6 [10.8 to 36.4] | 88.0 [48.6 to 127.5]
Statistical Analysis 1: Comparison: Sedation System vs Current Standard of Care; Test type: Superiority or Other; p = 0.028, ANOVA

2. Secondary Outcome: Duration of Deep Sedation/General Anesthesia
Description: Duration of Modified Observers Assessment of Alertness and Sedation (MOAA/S)score of 0 or 1 MOAA/S is a scale of numbers ranging from 0-5, 5 being defined as being awake or minimally sedatied, and 0 defined as being at the deepest level of sedation (general anethesia). The mean MOAA/S score was the sum of each subject's scores during the procedure divided by the number of non-missing scores.
Time Frame: From first dose until subject recovered from effects of sedation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sedation System | Current Standard of Care
Number analyzed (Participants) | 491 | 495
minutes | 0.1 (1.0) | 0.1 (1.1)

3. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction with Sedation Instrument (PSSI) is a scale measuring patient satisfactin with the sedation they received. This validated scale consists of 16 questions that are scored and converted to a 0-100 scale, where 100 represented the most satisfied.
Time Frame: 24-48 hours post sedation
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sedation System | Current Standard of Care
Number analyzed (Participants) | 392 | 397
Scores on a scale | 92.3 [91.0 to 93.5] | 89.7 [88.5 to 91.0]
Statistical Analysis 1: Comparison: Sedation System vs Current Standard of Care; Test type: Superiority or Other; p = 0.007, ANOVA

4. Secondary Outcome: Clinician Satisfaction
Description: Clinician Satisfaction with Sedation Instrument (CSSI) is a scale measuring the clinician satisfactin with the sedation they delivered. This validated scale consists of 16 questions that are scored and converted to a 0-100 scale, where 100 represented the most satisfied.
Time Frame: Post procedure
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sedation System | Current Standard of Care
Number analyzed (Participants) | 490 | 491
Scores on a scale | 92.2 [91.4 to 93.3] | 76.3 [74.8 to 77.8]
Statistical Analysis 1: Comparison: Sedation System vs Current Standard of Care; Test type: Superiority or Other; p < 0.001, ANOVA

5. Secondary Outcome: Recovery Time (From Sedation)
Description: Recovery time- time for patient to reach first of two consecutive MOAA/S of 5 from the time scope was removed.
Time Frame: from "scope out" until first of two consecutive MOAA/S scores of 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sedation System | Current Standard of Care
Number analyzed (Participants) | 463 | 465
minutes | 2.9 (2.4) | 6.5 (7.0)

ADVERSE EVENTS:
Arm/Group | Sedation System | Current Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/496 | 1/504
Other Adverse Events (participants affected / at risk) | 1/489 | 27/504
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedation System (N=496) | Current Standard of Care (N=504)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — hospitalization for abdominal pain, nausea and vomiting post colonoscopy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedation System (N=489) | Current Standard of Care (N=504)
Decreased Oxygen Saturation (Investigations) | 1 (1) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other